CLINICAL TRIAL: NCT02606981
Title: Evaluating Low-cost Automatic Water Disinfection Systems to Improve Water Quality and Child Health in Urban Bangladesh
Brief Title: Automatic Chlorination and Child Health in Urban Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Stephen P Luby, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 30456
Record Dates: First submitted 2015-10-20; First posted 2015-11-17 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diarrhea; Communicable Diseases
Keywords: Water treatment; Child growth; Enteric infection
MeSH Terms: conditions — Diarrhea; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorination (Experimental): Device: Water chlorination by the Flogenic Primary drinking water source will be outfitted with automatic dosing device supplied with chlorine tablets. The device is called the Flogenic.
  Interventions: Device: Water chlorination by the Flogenic
- Control (Placebo Comparator): Active control: Vitamin C dosing into water. Primary drinking water source will be outfitted with automatic dosing device supplied with vitamin C tablets. The device is not commercially available.
  Interventions: Device: Active control, vitamin C dosing into water

INTERVENTIONS:
Device: Water chlorination by the Flogenic — The chlorine doser delivers a constant amount of chlorine into water as it flows into a holding tank. The water is then piped to public and private taps.
  Other Names: Flogenic by Medentech
  Arms: Chlorination
Device: Active control, vitamin C dosing into water — The control group will receive a vitamin C dosing device that looks identical to the intervention chlorine doser installed in the holding tank that feeds their shared water access point.
  Other Names: Vitamin C dosing device (not commercially available)
  Arms: Control

SUMMARY:
Municipal water networks within industrialized countries typically rely on centralized treatment to manage piped water quality. Optimal water quality at the tap, however, requires well-maintained piped distribution networks, and performs best when piped systems are fully pressurized. In low-income cities such as Dhaka, water distribution networks are inadequately maintained and typically supply intermittent service; as such, they are vulnerable to recontamination during negative pressure events. Among populations accessing these types of improved water sources in urban settings (e.g. shared taps), it is unknown if consistent treatment to provide chlorinated water at the point of collection would have a significant health benefit. Furthermore, almost all previous studies of water treatment interventions in low-income countries have been unblinded with self-reported diarrhea as the main outcome, casting doubt that reported impacts of water disinfection on diarrhea are not due entirely to social desirability bias. Stanford University in collaboration with icddr,b will conduct a randomized evaluation to assess the impact on access to automatically chlorinated water on water quality and child health.

DETAILED DESCRIPTION:
Investigators will conduct a blinded cluster randomized controlled trial to evaluate the health and economic impacts of having access to automatically chlorinated water. The unit of randomization will be shared water points that typically serve 20-200 households. Shared water points connected to holding tanks compatible with the water treatment technology, and serving more than 4 households with at least one child under five, will be identified. Households accessing eligible water points as their primary drinking water source will be enrolled before installation of chlorine devices, and a baseline survey will be conducted of water quality, diarrhea prevalence, and health care expenditures. Following this baseline, households will be randomly assigned to control or treatment groups. The chlorination devices will be installed at the treatment group water points, while a doser containing vitamin C (and no chlorine), will be installed in the control group. The free chlorine dosing target will be below <1ppm to preserve blinding. All households will be surveyed every 2-3 months for a total follow up period of 14-16 months (5-7 survey rounds, budget permitting).

Objectives:

1. To evaluate the impact of an automated chlorination system on microbial stored drinking water quality, residual chlorine, user satisfaction, user perceptions of water taste and smell, under-five child diarrhea (longitudinal prevalence) compared to a control group.
2. Compare the marginal additional cost (per person served) of installing and maintaining an automated chlorination system integrated with the current water supply infrastructure in low-income areas of Dhaka.
3. Assess the impact of an automated chlorination system on hospital visits and health care expenditures.
4. To measure secondary outcomes of the impact of an automated chlorination system including under-five child weight-for-age (WAZ), under-five height-for-age (HAZ), as well as levels of C-reactive protein and immunoglobin G in serum samples collected from children under five (these are objective indicators of infection, such as repeat diarrheal episodes).

Analysis:

The primary analyses will be intent-to-treat (investigators will analyze differences in outcomes between the treatment and control groups, with groups defined by their random allocation). Investigators will also conduct a secondary analysis comparing outcomes between intervention and control, where the intervention group is defined as those households that had free chlorine residual detected in their stored drinking water (treated on the treated analysis).

ELIGIBILITY:
Inclusion Criteria:

* Households with at least one child under 60 months old
* Households using enrolled shared water point as primary drinking water source

Exclusion Criteria:

* Households with a private drinking water source

Note: New births and children under 60 months that migrate into compounds accessing the enrolled water points for drinking water will be enrolled into the study.

Max Age: 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1549 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Diarrhea longitudinal prevalence | Measured every 2-3 months for 16 months post baseline
  1-week recall period, case definition is 3 or more loose/watery bowel movements in 24 hours

SECONDARY OUTCOMES:
Weight-for-age-z-score | Measured every 2-3 months for 16 months post baseline
  Weight-for-age z-score among children under five years
Height-for-age-z-score | Measured at baseline and 16 months after baseline
  Height-for-age z-score among children under five
Respiratory illness longitudinal prevalence | Measured every 2-3 months for 16 months post baseline
  one week recall period, symptoms include congestion, cough, difficulty breathing
C-reactive protein | Measured at baseline and conclusion of study (16 months post baseline) among children under five
total immunoglobin G (IgG) | Measured at baseline and conclusion of study (16 months post baseline) among children under five
Prevalence and number of enteric pathogens | Measured 6-12 months after intervention delivery among children under five
Caregiver defined diarrhea | Measured every 2-3 months for 16 months post baseline
  1-week recall period, defined with local Bengali word for diarrhea

OTHER OUTCOMES:
Microbial water quality | Measured monthly among a subset of households, for 16 months post baseline
  Colony forming units of the fecal indicator bacteria, E. coli
Chlorine residual in household stored drinking water | Measured every 2-3 months for 16 months post baseline
  Free chlorine residual in ppm
health related treatment and associated cost | Measured every 2-3 months for 16 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Luby, MD, Principal Investigator — Stanford University; Amy Pickering, PhD, Study Director — Stanford University
Locations (1):
- Tongi and Dhaka Uddan, Tongi/Dhaka, Gazipur, Bangladesh

REFERENCES:
- [Derived] Pickering AJ, Crider Y, Sultana S, Swarthout J, Goddard FG, Anjerul Islam S, Sen S, Ayyagari R, Luby SP. Effect of in-line drinking water chlorination at the point of collection on child diarrhoea in urban Bangladesh: a double-blind, cluster-randomised controlled trial. Lancet Glob Health. 2019 Sep;7(9):e1247-e1256. doi: 10.1016/S2214-109X(19)30315-8. PMID 31402005